CLINICAL TRIAL: NCT04484714
Title: Feasibility of a Virtually Supported Home-Based Resistance and Aerobic Exercise Program for Cancer Survivors With Multiple Myeloma
Brief Title: Virtual Exercise for Multiple Myeloma
Acronym: MY-PROGRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-20-0201
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Multiple Myeloma
Keywords: exercise; pilot; feasibility
MeSH Terms: conditions — Multiple Myeloma; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single group before and after
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioural: Exercise (Experimental): Participants will take part in a twelve week resistance and aerobic exercise program twice per week delivered virtually.
  Exercise sessions will include a combination of aerobic, resistance, balance, and flexibility exercises
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will participate in a 12-week virtually supported home-based aerobic and resistance exercise program, twice weekly using the Heal-Me application. Sessions will be completed as virtual live classes or supported follow-along independent home workouts. Sessions will progress in duration and difficulty over the course of the program, aiming to have participants meet the 2019 Exercise Guidelines for Cancer Survivors by the end of the program. Each session will include aerobic exercise (i.e. walking, cycling, or cardio circuit), and a full-body resistance training routine using free weights, body weight exercises, and/or bands, followed by balance and stretching exercises.

SUMMARY:
The primary objective of this pilot study is to determine the safety and feasibility a 12-week virtually supported home-based aerobic and resistance exercise program progressing cancer survivors with Multiple Myeloma to meet standards identified in the 2019 Exercise Guidelines for Cancer Survivors.

The protocol will be measuring recruitment, adherence, completion, cost tracking, as well as fitness and quality of life outcomes. The study will be a single-group prospective before and after study that will help inform a future larger-scale project. We will aim to recruit 25 participants.

The Health Research Ethics Board of Alberta Cancer Committee will approve this study. Participants will participate in a combined resistance and aerobic exercise program biweekly for 12 weeks. Exercise sessions will be supported and progressive in nature, between 40 and 75 minutes each.

Analyses: fitness testing and quality of life scales will be administered before and after the intervention. Scores will be compared to evaluate changes over the course of the intervention. Safety and feasibility information will be collected throughout the study and evaluated to determine program feasibility. Program satisfaction will be evaluated using a satisfaction survey.

DETAILED DESCRIPTION:
Multiple myeloma (MM), a cancer of the plasma cells in bone marrow, is associated with osteolytic bone destruction, leading to deformities, chronic pain, reduced mobility and functioning, fatigue, and risk of fracture. Although incurable, newly developed therapies are extending survival, but some with significant side-effects. Patients may be living longer but with lasting, debilitating side-effects.

Exercise has been proposed as a way to optimize patient function and quality of life in the face of lasting symptom burden. However, current evidence-informed exercise guidelines for cancer survivors may not be appropriate for those with bone fragility, including those with MM, as they are based on findings from studies in breast and prostate cancers. In MM specifically, the literature presents mixed results, and several studies have limited generalizability, reproducibility, or were underdosed.

The main objective of this study is to determine the safety and feasibility of a 12-week virtually supported home-based aerobic and resistance exercise program that aims to progress individuals to the 2019 Exercise Guidelines for Cancer Survivors in a sample of cancer survivors with multiple myeloma, as defined by:

* Recruitment rate: ≥ 21 participants consenting to the study over a 7-month recruitment period (primary endpoint)
* Completion rate: ≥ 80% of participants consenting to the study complete the 12-week assessment
* Safety: no increase in the rate of bony events above those estimated to occur in the target population
* Adherence: average completion of ≥ 75% of the exercise prescription amongst participants

We will aim to recruit 25 participants from clinics at the local cancer hospital, the local disease-group support society, and from the currently accruing Alberta Cancer Exercise program. Subjects will be screened for eligibility and if they meet all eligibility criteria, an information letter of the study will be provided, and they will be asked to contact the investigators if interested in taking part in the study. All participants will be required to provide written informed consent as per the Health Research Ethics Board of Alberta: Cancer Committee (HREBA).

Participants will participate in a 12-week virtually supported home-based aerobic and resistance exercise program, twice weekly using the Heal-Me application. Sessions will be completed as virtual live classes or supported follow-along independent home workouts. Sessions will progress in duration and difficulty over the course of the program, aiming to have participants meet the 2019 Exercise Guidelines for Cancer Survivors by the end of the program. Each session will include aerobic exercise (i.e. walking, cycling, or cardio circuit), and a full-body resistance training routine using free weights, body weight exercises, and/or bands, followed by balance and stretching exercises.

Analyses: Demographic and medical information will be presented using median and range and percentage for interval and nominal data, respectively. Descriptive statistics (mean ± SD and frequencies) will be used to report safety and feasibility measures. Adherence will be tracked as the percentage of total training load prescribed that was actually completed. Wilcoxon Signed Rank Tests will be used to compare and pre- and post-intervention fitness assessment and quality of life scores. All analyses will be conducted using Stata/MP (version 13.0, StataCorp LLC, College Station, TX), with alpha set to 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Diagnosis of multiple myeloma
3. In one of the following three treatment categories:

   * Transplant ineligible patients, currently in first line treatment
   * Transplant eligible patients, sufficiently recovered from transplantation (>3 months following transplantation)
   * Patients with relapsed/recurrent myeloma with either 1-3 prior lines of treatment or 4+ prior lines
4. Able to provide informed written consent in English
5. Approved for physical activity participation by their oncologist and cleared for physical activity by the Certified Exercise Physiologist on the PAR-Q+

Exclusion Criteria:

1. Unstable cardiac/metabolic condition that would be deemed unsafe to exercise
2. Severe anemia
3. Spinal instability requiring surgical intervention
4. AL amyloidosis, solitary plasmacytoma, or Waldenstrom macroglobulinemia
5. Too frail to participate in home exercise, as determine by baseline physical assessment (i.e., unable to complete a single sit-to-stand or balance on one foot for ≥ 3 seconds).
6. Inability to provide consent
7. Inability to commit to, and/or comply with the intervention due to personal reasons (e.g. vacation planned during the intervention period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility (Adherence) | 12 weeks
  The percentage of total exercise dose prescribed that was actually completed (%)

SECONDARY OUTCOMES:
Feasibility (Recruitment rate) | 7 months
  The number of participants recruited per month over the recruitment period and the proportion of patients who participate in the study, out of the total number of eligible patients
Feasibility (Completion rate) | 12 weeks
  The number of participants who completed the program and follow-up assessment out of the number of participants who consented to the study
Feasibility (Safety) | 12 weeks
  The number of adverse events reported by the participants during program participation, including the 12-week program and fitness assessments

OTHER OUTCOMES:
Home-based Stepping Test | Change from baseline to 12 weeks
  Change in 2-minute stepping test (number of steps)
Shoulder flexibility | Change from baseline to 12 weeks
  Change in active shoulder flexion range of motion (degrees)
Lower Body Flexibility | Change from baseline to 12 weeks
  Change in sit-and-reach test (cm)
Leg Strength | Change from baseline to 12 weeks
  Change in 30-second sit-to-stand (number of repetitions)
Balance | Change from baseline to 12 weeks
  Change in one legged stance test (seconds
Balance Confidence | Change from baseline to 12 weeks
  Activities-specific Balance Confidence (ABC) scale (score)
Upper Extremity Function | Change from baseline to 12 weeks
  Change in Upper Extremity Functional Index (score)
Lower Extremity Function | Change from baseline to 12 weeks
  Change in Lower Extremity Functional Scale (score)
Cancer-Specific Quality of Life | Change from baseline to 12 weeks
  Change in Functional Assessment of Cancer Therapy General, Multiple Myeloma, and Bone Pain Scales (score)
Fatigue | Change from baseline to 12 weeks
  Change in FACIT-Fatigue Subscale (score)
Six-minute walk test (optional) | Change from baseline to 12 weeks
  Six-minute walk test distance (metres)
Upper Extremity Grip Strength (optional) | Change from baseline to 12 weeks
  Hand-grip dynamometry (kg)
Upper extremity strength (optional) | Change from baseline to 12 weeks
  One repetition maximum bench press (kg)
Lower extremity strength (optional) | Change from baseline to 12 weeks
  One repetition maximum leg press (kg)
Core Endurance (optional) | Change from baseline to 12 weeks
  Plank hold (seconds)
Fall risk (optional) | Change from baseline to 12 weeks
  Three-metre backwards walk test (seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta/ Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
No plan in place at this time